CLINICAL TRIAL: NCT04081753
Title: Remote Outpatient Temperature Monitoring for Early Detection of Febrile Neutropenia After Chemotherapy
Acronym: REMEDY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: University of Georgia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1464778
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-07

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: HiDAC; Neutropenia; Fever; AML; Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neutropenia; Fever; Leukemia

STUDY DESIGN:
Intervention Model Description: Interventional group will be compared with historic group of patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TMD Group (Experimental): Temperature Monitoring Device Group - The interventional group, who will be given the temperature monitoring device and will be monitored remotely.
  Interventions: Device: Remote monitoring of temperature
- Historic cohort Group (No Intervention): Historic cohort group will be enrolled from medical record

INTERVENTIONS:
Device: Remote monitoring of temperature — The patient will be set up with a remote monitoring device for temperature recording and the temperature will monitored remotely
  Arms: TMD Group

SUMMARY:
Febrile neutropenic patients are at high risk for developing sepsis and other infections which often necessitates acute admission to the Intensive Care Unit (ICU) and are associated with high mortality. Neutropenic fever is a medical emergency and early detection of fever allows for prompt infectious work up. In this study, the investigators will collect pilot data from outpatients utilizing a remote outpatient continuous temperature monitoring device to compare the incidence of ICU admission and severe sepsis to historical data for prior patients who did not receive at home monitoring device.

ELIGIBILITY:
Inclusion Criteria:

Patients who have acute myeloid leukemia (AML) and are candidates for consolidation chemotherapy with high dose cytarabine (HiDAC) after successful remission induction chemotherapy

* Both male and female
* Age 18 years and older

Exclusion Criteria:

Patients who have already developed febrile neutropenia during their hospitalization for their consolidative cycle of chemotherapy will not be eligible for monitoring for that cycle; however, these patients will be able to participate in subsequent cycle if they do not develop febrile neutropenia during their subsequent HiDAC hospitalization.

• If a patient is admitted to the hospital between cycles of chemotherapy for reasons other than febrile neutropenia or its sequelae, they will be taken off study for that cycle and data not collected while they are admitted

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change ICU admission | 1 month
  The interventional group will have changed in the number of ICU admission.
Change incidence of sepsis in interventional group | 1 month
  The interventional group will have changed rate of sepsis incidence.

CONTACTS AND LOCATIONS:
Overall Officials: Locke J. Bryan, MD, Principal Investigator — Augusta University
Locations (1):
- Augusta University Medical Center, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
This study result will be used for service improvement of patient of the Augusta University Medical Center

REFERENCES:
- [Background] Pathak R, Giri S, Aryal MR, Karmacharya P, Bhatt VR, Martin MG. Mortality, length of stay, and health care costs of febrile neutropenia-related hospitalizations among patients with breast cancer in the United States. Support Care Cancer. 2015 Mar;23(3):615-7. doi: 10.1007/s00520-014-2553-0. Epub 2015 Jan 4. PMID 25556610
- [Background] Saini L, Rostein C, Atenafu EG, Brandwein JM. Ambulatory consolidation chemotherapy for acute myeloid leukemia with antibacterial prophylaxis is associated with frequent bacteremia and the emergence of fluoroquinolone resistant E. Coli. BMC Infect Dis. 2013 Jun 22;13:284. doi: 10.1186/1471-2334-13-284. PMID 23800256
- [Background] van Vliet M, Donnelly JP, Potting CM, Blijlevens NM. Continuous non-invasive monitoring of the skin temperature of HSCT recipients. Support Care Cancer. 2010 Jan;18(1):37-42. doi: 10.1007/s00520-009-0627-1. Epub 2009 Apr 25. PMID 19396473
- [Background] Freifeld AG, Bow EJ, Sepkowitz KA, Boeckh MJ, Ito JI, Mullen CA, Raad II, Rolston KV, Young JA, Wingard JR; Infectious Diseases Society of America. Clinical practice guideline for the use of antimicrobial agents in neutropenic patients with cancer: 2010 update by the infectious diseases society of america. Clin Infect Dis. 2011 Feb 15;52(4):e56-93. doi: 10.1093/cid/cir073. PMID 21258094
- [Background] Taplitz RA, Kennedy EB, Bow EJ, Crews J, Gleason C, Hawley DK, Langston AA, Nastoupil LJ, Rajotte M, Rolston K, Strasfeld L, Flowers CR. Outpatient Management of Fever and Neutropenia in Adults Treated for Malignancy: American Society of Clinical Oncology and Infectious Diseases Society of America Clinical Practice Guideline Update. J Clin Oncol. 2018 May 10;36(14):1443-1453. doi: 10.1200/JCO.2017.77.6211. Epub 2018 Feb 20. PMID 29461916